CLINICAL TRIAL: NCT07038486
Title: The Impact of a Digital System on the Monitoring and Self-management of Non-motor Symptoms in People With Parkinson's
Brief Title: Patient Engagement Investigation of NMS Assist
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Principal Investigator, Edward Meinert, Professor of Digital Health and Clinical Artificial Intelligence, Newcastle University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202425 16 Caroll; H-2101 (Other Grant/Funding Number: Parkinson's UK)
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Self-management; mhealth; mobile apps; telemedicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NMS Assist (Experimental): NMS Assist provides a system of linking PwP, CPs, and healthcare providers (HCPs) to monitor and empower self-management of non-motor symptoms through the use of a mobile app and web portal.
  Interventions: Device: NMS Assist

INTERVENTIONS:
Device: NMS Assist — The system enables people with Parkinson's and their care partners to complete questionnaires about symptoms and burden and share that information with their care team. They can also access self-help resources and materials about managing non-motor symptoms. Healthcare providers have a dashboard that flags any worsening symptoms or discrepancies between PwP and CP reports, enabling their to prioritise care and quickly see the status of their patients. The system also enables PwP or CPs to request healthcare contact.

SUMMARY:
Parkinson's can cause a wide range of non-motor symptoms (NMS), including pain and problems with mental health, memory and sleep. These affect the quality of life of people with Parkinson's (PwP) and their care partners (CP). If these issues are not recognised and managed quickly, they can result in escalating problems. Many PwP are unsure of the extent and variety of the NMS and how simple adjustments at home could improve them. We have developed a digital system to help PwP monitor their non-motor symptoms and develop skills to self-manage them.

Such a tool needs to be simple to use, safe and effective. We will ask 30 PwP and CPs to use the digital tool for 6 months, and we will monitor how they use the tool. PwP and CPs will be asked if they feel more knowledgeable and confident to manage their own symptoms whilst being better able to discuss a problem with their healthcare professional.

A smaller group of participants will discuss their experiences in more detail to help pinpoint aspects that work well and those needing adjustment and development.

It is thought that the use of this system will result in improved quality of life and increased knowledge and confidence for managing symptoms while safely reducing the time spent by healthcare professionals on manageable non-motor symptoms.

ELIGIBILITY:
Inclusion Criteria: Individuals will be eligible if they meet the following inclusion criteria:

All:

* Age 18 years or over
* Have compatible smartphone/data access (access to a digital device is a necessary prerequisite of system use, and the formative usability study had success in recruiting participants with varying levels of experience with smartphones)
* Be fluent in English
* Able and willing to provide informed consent
* Able and willing to comply with intervention requirements

For clinically diagnosed people with Parkinson's (PwP) (ICD-10-CM G20):

* Not resident in a care home or nursing home
* Ambulant
* Interested in monitoring and managing their NMS

For CPs:

- Be caring for a clinically diagnosed PwP (ICD-10-CM G20) who is participating in the study

Exclusion Criteria: Participants will be ineligible for the study if they meet any of the following exclusion criteria:

All:

* Previous involvement in the development or testing of the digital system
* In a dependent/unequal relationship with the research or care teams or any PPI representatives

PwP:

* Secondary cause of Parkinsonism
* Significant cognitive impairment or a diagnosis of Parkinson's disease dementia
* Significant comorbidity, which, in the opinion of the chief investigator, would preclude safe participation in the study or protocol compliance
* A life expectancy of <6 months
* Living in residential care facilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | Assessed throughout the 6-month study duration
  The primary outcome will be assessed using a composite of variables: recruitment, retention, system uptime, adherence/engagement, technical issues, and a review of the health and well-being outcomes (secondary outcomes).
  Adherence/engagement will be measured using system use data (trend of use over time). This will be supplemented with semi-structured interviews and a user engagement questionnaire to gain a better understanding of users' experience engaging with the intervention and the recommended behaviours. Technical issues will be identified through system use data (including logs of complaints made by participants during the intervention delivery period) as well as asking participants about any technical issues encountered during the semistructured interviews. Product complaints will be collected through feedback recorded via the platform, collected at study assessment points or manually provided via email throughout the study duration.

SECONDARY OUTCOMES:
Presence of non-motor symptoms | Measured monthly for 6 months
  Measured using the Non-Motor Symptoms Questionnaire (NMSQ), patients tick 'yes' or 'no' for each symptom listed
Patient (and care partner) activation | Assessed monthly for 6 months
  Patient Activation Measure (and caregiver version) will be used to evaluate their confidence, knowledge, and skills at non-motor symptom self-management
Frequency and severity of non-motor symptoms | Measured at baseline, 3, and 6 months
  Measured using the Movement Disorder Society Non-Motor Symptoms Scale (MDS-NMS), where higher scores indicate greater frequency and/or severity
Long-form self-assessment of functioning and well-being related to Parkinson's disease | Measured at baseline, 3, and 6 months
  Measured using the long-form Parkinson's Disease Questionnaire PDQ-39, patients indicate the frequency with which they experience certain issues
Short-form self-assessment of functioning and well-being related to Parkinson's disease | Measured monthly for 6 months
  Measured using the short-form Parkinson's Disease Questionnaire (PDQ-8), patients indicate the frequency with which they experience certain issues
Carer well-being and quality of life | Measured monthly for 6 months
  Measured using the Parkinson Disease Questionnaire for care partners; care partners indicate the frequency with which they experience certain issues
Health status | Measured at baseline, 3, and 6 months
  Measured using the EQ-5D-5L; higher scores on the EQ-5D-5L descriptive system indicate worse health problems in the specific dimension whereas a high score in the EQ VAS indicates better health on the day of the questionnaire
Adverse events | Throughout the 6-month study period
  Adverse event reporting
Healthcare contacts | Throughout the 6-month study period
  Number of PwP-initiated contacts with healthcare team (through the 'request healthcare contact' feature) recorded by the system
Quantitative usability | 3 and 6 months
  Using the mHealth app usability questionnaire (MAUQ) with higher scores indicating better usability
Acceptability | 3 and 6 months
  Acceptability and usability feedback from semi-structured interviews
Costs will be conducted, in conjunction with an adaptation of Client Service Receipt Inventory (CSRI) | Throughout 6 months
  Cost analysis will be conducted, in conjunction with an adaptation of Client Service Receipt Inventory (CSRI) for Parkinson's disease. The scale will be administered at 3 and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Newcastle University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data belongs to the study sponsor (Newcastle University) and deidentified data will be made available in line with the data sharing policy developed with Parkinson's UK and PPI representatives.